CLINICAL TRIAL: NCT02613572
Title: Evaluation of Lipoic Acid as a Treatment for Geographic Atrophy Secondary to Age-Related Macular Degeneration (AMD): Phase I- Tolerability Study and Phase II Pilot- Determine the Effects of ALA on the Progression of Geographic Atrophy (GA) in Patients With Age-related Macular Degeneration (AMD).
Brief Title: Alpha Lipoic Acid in Geographic Atrophy
Acronym: ALA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 822310; 822311 (Other: University of Pennsylvania, Coordinating IRB); 201604726 (Other: University of Iowa, IRB)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- alpha lipoic acid (ALA) 600mg once daily x 5 days (Experimental): All 15 patients recruited to the Phase I part will take escalating doses of alpha lipoic acid (ALA) open label. Each enrolled subject will take 600 mg of oral ALA once daily with a meal for 5 days. If well-tolerated, each subject will then take 800 mg of oral ALA once daily with a meal for 5 additional days. If 800 mg of oral ALA is well-tolerated, then subjects will then take 1200 mg of oral ALA once daily with a meal for 5 days.
  Interventions: Drug: alpha lipoic acid
- alpha lipoic acid 800mg (Experimental): once daily with meal x 5 days
  Interventions: Drug: alpha lipoic acid
- alpha lipoic acid 1200mg (Experimental): once daily x 5 days
  Interventions: Drug: alpha lipoic acid
- Placebo 600mg (Placebo Comparator): All 50 subjects in Phase II will be double blinded and randomized to either placebo or ALA. Each will take one 600mg capsule of ALA (or placebo) once daily with a meal for 2 weeks and then increase to two 600 mg capsules of ALA (or placebo) once daily with a meal for the
  Interventions: Drug: Placebo
- ALA 600 mg (Experimental): once daily with a meal for 2 weeks
  Interventions: Drug: alpha lipoic acid
- Placebo 1200mg (Placebo Comparator): Two 600mg capsules once daily with a meal for the entire remainder of the 18 month period of the study
  Interventions: Drug: Placebo
- ALA 1200mg (Experimental): Two 600mg capsules once daily with a meal for the entire remainder of the 18 month period of the study
  Interventions: Drug: alpha lipoic acid

INTERVENTIONS:
Drug: alpha lipoic acid
  Other Names: thioctic acid
  Arms: ALA 1200mg; ALA 600 mg; alpha lipoic acid (ALA) 600mg once daily x 5 days; alpha lipoic acid 1200mg; alpha lipoic acid 800mg
Drug: Placebo
  Arms: Placebo 1200mg; Placebo 600mg

SUMMARY:
Because of its iron-chelating and antioxidant properties, alpha lipoic acid may be a treatment for geographic atrophy (GA) secondary to age-related macular degeneration. There is ample published data about the safety and pharmacokinetics of alpha lipoic acid in adults. However, there is not much data on the safety and tolerability of higher doses of alpha lipoic acid in the elderly population. The purpose of Phase I of this protocol is to determine if there are safety/tolerability concerns seen when higher doses of alpha lipoic acid are taken by subjects 65 years of age or older.

The objective of Phase 2 of this protocol is to determine the effects of ALA on the progression of GA in subjects with AMD. The central hypothesis, based on the existing literature, is that oral ALA reduces the rate of enlargement of GA in AMD subjects. The rationale is that the antioxidant and iron chelating effects of ALA will slow down one of the major pathways responsible for GA progression.

DETAILED DESCRIPTION:
Phase I (Apr 2016 completed): 15 subjects, 65 years of age or older will take alpha lipoic acid on the following schedule:

600 mg once daily with a meal for 5 days. If tolerated, then the subject will then take 800 mg once daily with a meal for 5 days.

If tolerated, then the subject will then take 1200 mg once daily with a meal for 5 days.

Phase II: Randomized, double-blind placebo controlled pilot trial. Upon the completion of the dose tolerability test, we plan to enroll 50 subjects into a randomized, double-blind, placebo-controlled trial. Subjects will be randomized (1:1) into one of two study arms: placebo capsules and ALA 1200 mg orally once daily, assuming that 1200 mg is well tolerated by subjects in Phase 1. If 1200 mg is not well-tolerated based on Phase 1 data, then the highest tolerable dose will be used. Four clinical sites are planned and the enrollment period is estimated to be 6 months. The primary endpoint is the mean rate of change of the area of GA in the study eye from baseline to 18 months as evaluated by fundus autofluorescence. Subjects will have a refracted electronic visual acuity and dilated exam at baseline, 6 months, 12 months, and 18 months. The study will be conducted on an outpatient basis and study visits will last approximately 2-3 hours. Two weeks after the 18 months study visit, the subject will be contacted to share with the investigators adverse events that developed after completing the 18 month visit. The Investigator shall ensure each subject has a follow-up eye exam scheduled within 6 months.

ELIGIBILITY:
Phase I

Inclusion Criteria:

* Ages 65-90
* Female participants must be menopausal. Male participants are required to use contraception.
* Able to give informed consent
* For the study duration (15 days), the subject must remain in the country, remain within 4 hours of travel time (by car or airplane), have access to medical care if needed, and provide contact information so the subject can be reached as needed.

Exclusion Criteria:

* Blood Pressure greater than 190/100 at the baseline visit
* Pulse greater than 100 at the baseline visit
* Acute and ongoing systemic infection
* History of dementia
* Participant has a condition that, in the opinion of the investigator, gives them an unstable medical status.
* Participant has geographic atrophy and the investigator believes the participant is a candidate for enrollment into the planned Phase 2 trial for geographic atrophy.

Phase II

Inclusion Criteria

* Age 55-90
* Diagnosis of geographic atrophy from age-related macular degeneration in the study eye. The largest geographic atrophy (GA) lesion must be a minimum of 0.5 optic disk area (DA) (1.25 mm2) and no more than 6 DA in size (15.0 mm2). GA is defined as one or more well-defined, usually more or less circular patches of loss of the retinal pigment epithelium (RPE), typically with exposure of underlying choroidal blood vessels. If the GA is multifocal and the largest lesion is < 0.5 DA, then there should be at least 3 lesions ≥ 250 microns in greatest linear diameter.
* Best-Corrected Visual Acuity (BCVA) between 20/20 and 20/400 in the study eye.
* Female participants must be menopausal. Male participants are required to use contraception and cannot donate sperm during study participation.
* Presence of hyperfluorescence at the edge of GA on autofluorescence imaging.
* Ability to give informed consent.
* If a subject has two eligible eyes, then both eyes can be enrolled into the study.
* Subject must have mailed back the medication bottle after the 10 day run-in phase, demonstrating that they have taken ≥ 80% of the capsules.

Exclusion Criteria

* Evidence of ocular disease other than AMD in the study eye that may confound the study outcomes (e.g., History of myopic degeneration, choroidal neovascularization, central serous chorioretinopathy, severe diabetic retinopathy, uveitis, vitelliform dystrophy, or macular edema).
* Presence of geographic atrophy that is already touching clearly defined beta peripapillary atrophy or is already touching the optic disc. Beta peripapillary atrophy is defined as peripapillary atrophy in which either the sclera or choroidal vessels are clearly visible.
* Any history of intravitreal injection in the study eye for AMD or choroidal neovascularization.

However, if a subject develops choroidal neovascularization in the study eye during the study, then the subject will receive the standard of care intravitreal injection treatments per the investigator. The subject will continue to stay in the study. Treatment of choroidal neovascularization (CNV) or other diseases in the non-study eye is at the investigator's discretion.

* History of intravitreal injection of any agent (e.g., triamcinolone) other than anti-VEGF (vascular endothelial growth factor) in the study eye within the last four months prior to study enrollment.
* History of laser treatment (including photodynamic therapy) to the macula for the study eye.
* History of intraocular surgery within 90 days. for the study eye.
* History of anterior segment laser (laser peripheral iridotomy, laser to trabecular meshwork, YAG capsulotomy) within 90 days for the study eye.
* Media opacity (corneal scar, cataract) that would prevent adequate fundus imaging for the study eye.
* Any history of participation in another therapeutic clinical trial for GA.
* Participation currently or within the past 30 days in another therapeutic clinical trial in which a systemic or ocular study medication is received by the subject.
* GA in the study eye due to a cause other than AMD
* History of prior use of ALA.
* AREDS (Age Related Eye Disease Study) vitamins taken at standard doses are not considered an exclusion criterion. Taking a standard multivitamin is not considered an exclusion criterion. However, the multivitamin should not contain alpha lipoic acid (also known as thioctic acid).
* Taking antioxidant supplements other than a standard multivitamin (such as bilberry, vitamin C that is not part of a multivitamin or taken at higher doses than the AREDS formula, vitamin E that is not part of a multivitamin or taken at higher doses than the AREDS formula, or other similar antioxidants) within one month of enrollment is an exclusion criteria; these patients should discontinue the antioxidant supplement one month before enrollment in order to participate. Taking a supplement that has antioxidant potential that is recommended by a physician as standard-of-care medical management is not an exclusion criterion.).
* Participant has a condition that, in the opinion of the investigator, would preclude participation in the study for 18 months (e.g., unstable medical status including blood pressure and glycemic control, unstable psychiatric history, moving and not able to return for all planned study visits).
* History of a formal diagnosis of dementia by a neurologist.
* History of gastric ulcer within the past 5 years.
* History of irritable bowel syndrome within the past 5 years.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11; Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Kim, MD, Study Chair — University of Pennsylvania
Locations (5):
- United States (5):
  - University of Iowa Hospitals and Clinics, Department of Ophthalmology & Visual Sciences, Iowa City, Iowa
  - NJ Retina, Teaneck, New Jersey
  - Oregon Regina. LLP, Eugene, Oregon
  - Retina Northwest, P.C., Portland, Oregon
  - Scheie Eye Institute of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Sarezky D, Raquib AR, Dunaief JL, Kim BJ. Tolerability in the elderly population of high-dose alpha lipoic acid: a potential antioxidant therapy for the eye. Clin Ophthalmol. 2016 Sep 29;10:1899-1903. doi: 10.2147/OPTH.S115900. eCollection 2016. PMID 27729766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I: 15 subjects took escalating ALA doses (600mg, 800mg, 1200mg). 1 subject withdrew after 800mg due to wanting to delay start of 1200mg dose beyond planned completion date.
  Phase II: 52 subjects randomized to placebo or 1200mg ALA. 1 subject died due to unrelated event and was replaced in study; thus, 53 total subjects were enrolled.
Groups:
- Alpha Lipoic Acid (ALA) 600, 800, 1200 mg: Phase I: All subjects recruited to the Phase I part will take escalating doses of alpha lipoic acid (ALA) open label. Each enrolled subject will take 600 mg of oral ALA once daily with a meal for 5 days. If well-tolerated, each subject will then take 800 mg of oral ALA once daily with a meal for 5 additional days. If 800 mg of oral ALA is well-tolerated, then subjects will then take 1200 mg of oral ALA once daily with a meal for 5 days.
- Placebo 1200mg; Alpha Lipoic Acid (ALA) 1200mg: Phase II: All subjects in Phase II will be double blinded and randomized to either placebo or ALA. Each will take one 600 mg capsule of ALA (or placebo) once daily with a meal for 2 weeks and then increase to two 600 mg capsules of ALA (or placebo) once daily with a meal for the entire remainder of the 18 month period of the study.
Period: Phase I: Tolerability, 600, 800, 1200 mg
Arm/Group | Alpha Lipoic Acid (ALA) 600, 800, 1200 mg | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Started | 15 | 0 | 0
600 mg | 15 | 0 | 0
800 mg | 15 | 0 | 0
1200 mg | 14 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Phase II: Double-Blind Rand Plac Control
Arm/Group | Alpha Lipoic Acid (ALA) 600, 800, 1200 mg | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Started | 0 | 27 | 26
Completed | 0 | 26 | 26
Not Completed | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alpha Lipoic Acid (ALA) 600, 800 &1200 mg: Phase I: All subjects recruited to the Phase I part will take escalating doses of alpha lipoic acid (ALA) open label. Each enrolled subject will take 600 mg of oral ALA once daily with a meal for 5 days. If well-tolerated, each subject will then take 800 mg of oral ALA once daily with a meal for 5 additional days. If 800 mg of oral ALA is well-tolerated, then subjects will then take 1200 mg of oral ALA once daily with a meal for 5 days.
- Total: Total of all reporting groups
Arm/Group | Alpha Lipoic Acid (ALA) 600, 800 &1200 mg | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg | Total
Number analyzed (Participants) | 15 | 27 | 26 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (3.3) | 79.0 (7.0) | 80.6 (6.5) | 77.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 18 | 44
  Male | 5 | 11 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 12 | 26 | 24 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 27 | 26 | 68
Bilateral Geographic Atrophy [Count of Participants; unit: Participants] — Population: Phase I (Alpha Lipoic Acid (ALA) 600, 800 &1200 mg) subjects did not have their eyes measured for Bilateral Geographic Atrophy, which is why no patients are included in the count of participants for this baseline measure.
  Participants
    Yes: number analyzed (Participants) | 0 | 27 | 26 | 53
    Yes | 0 | 24 | 23 | 47
    No: number analyzed (Participants) | 0 | 27 | 26 | 53
    No | 0 | 3 | 3 | 6
Geographic Atrophy Lipoic Acid Study (GALA) Eligible Eyes [Count of Participants; unit: Participants] — Population: Phase I (Alpha Lipoic Acid (ALA) 600, 800 &1200 mg) subjects did not have their eyes measured for Geographic Atrophy Lipoic Acid Study (GALA) Eligible Eyes, which is why no patients are included in the count of participants for this baseline measure.
  Participants
    Unilateral: number analyzed (Participants) | 0 | 27 | 26 | 53
    Unilateral | 0 | 17 | 16 | 33
    Bilateral: number analyzed (Participants) | 0 | 27 | 26 | 53
    Bilateral | 0 | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Percentage of Participants With Adverse Events
Description: The percent of adverse events that develop will be stratified by the alpha lipoic acid dose.
Time Frame: 15 days
Population: Phase I: 15 subjects took escalating ALA doses (600mg, 800mg, 1200mg). 1 subject withdrew after 800mg due to wanting to delay start of 1200mg dose beyond planned completion date.
Measure: Count of Participants; unit: Participants
Groups:
- Alpha Lipoic Acid (ALA) 600 mg; Alpha Lipoic Acid (ALA) 800 mg; Alpha Lipoic Acid (ALA) 1200 mg: Phase I: All subjects recruited to the Phase I part will take escalating doses of alpha lipoic acid (ALA) open label. Each enrolled subject will take 600 mg of oral ALA once daily with a meal for 5 days. If well-tolerated, each subject will then take 800 mg of oral ALA once daily with a meal for 5 additional days. If 800 mg of oral ALA is well-tolerated, then subjects will then take 1200 mg of oral ALA once daily with a meal for 5 days.
Arm/Group | Alpha Lipoic Acid (ALA) 600 mg | Alpha Lipoic Acid (ALA) 800 mg | Alpha Lipoic Acid (ALA) 1200 mg
Number analyzed (Participants) | 15 | 15 | 14
Participants | 11 | 10 | 10
Statistical Analysis 1: Comparison: Alpha Lipoic Acid (ALA) 600 mg vs Alpha Lipoic Acid (ALA) 800 mg vs Alpha Lipoic Acid (ALA) 1200 mg; Test type: Superiority; p = 1.00, Fisher Exact

2. Primary Outcome: Phase II: Mean Annual Growth of Geographic Atrophy (Fundus Autofluorescence) - Total Area of Geographic Atrophy (mm2) - Unadjusted
Description: The rate of change over time in area of Geographic Atrophy (GA) in the study eye. This is determined by masked grading of Fundus Autofluorescence by an image reading center, in participants randomized to placebo or 1200 mg once daily of ALA. The values represent the annualized change from baseline to 18 months. Mean annual geographic atrophy growth rate was calculated by taking the total atrophy area at 18 months minus the baseline area. This value was then divided by 18 months and then multiplied by 12 months to get the annual growth rate. Timepoints for the study were baseline, 0, 6, 12, and 18 months. The baseline and 18 month timepoints were used for the annualized calculations as noted below.
Time Frame: 18 months
Population: Phase II: 52 subjects randomized to placebo or 1200mg ALA. 1 subject died due to unrelated event and was replaced in study; thus, 53 total subjects were enrolled, but 52 subjects were analyzed in this outcome.
Measure: Mean (Standard Deviation); unit: mm^2/year
Arm/Group | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Number analyzed (Participants) | 26 | 26
mm^2/year | 1.21 (0.13) | 1.71 (0.13)
Statistical Analysis 1: Comparison: Placebo 1200mg vs Alpha Lipoic Acid (ALA) 1200mg; Test type: Superiority; p = 0.009, Mixed Models Analysis

3. Primary Outcome: Phase II: Mean Annual Growth of Geographic Atrophy (Fundus Autofluorescence) - Total Area of GA (mm2) - Adjusted
Description: as for outcome 2
Time Frame: 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2/year
Arm/Group | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Number analyzed (Participants) | 26 | 26
mm^2/year | 1.29 (0.23) | 1.63 (0.28)
Statistical Analysis 1: Comparison: Placebo 1200mg vs Alpha Lipoic Acid (ALA) 1200mg; Test type: Superiority; p = 0.09, Mixed Models Analysis

4. Primary Outcome: Phase II: Mean Annual Growth of Geographic Atrophy (Fundus Autofluorescence) - Square Root of Area of GA (mm) - Unadjusted
Description: The rate of change over time in area of Geographic Atrophy (GA) in the study eye. This is determined by masked grading of Fundus Autofluorescence (FAF) by an image reading center, in participants randomized to placebo or 1200 mg once daily of ALA. The values represent the annualized change from baseline to 18 months. Mean annual geographic atrophy growth rate was calculated by taking the total atrophy area at 18 months minus the baseline area. This value was then divided by 18 months and then multiplied by 12 months to get the annual growth rate. For square root transformed data, the square root of area was used. Timepoints for the study were baseline, 0, 6, 12, and 18 months. The baseline and 18 month timepoints were used for the annualized calculations as noted below.
Time Frame: 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Number analyzed (Participants) | 26 | 26
mm/year | 0.28 (0.02) | 0.31 (0.02)
Statistical Analysis 1: Comparison: Placebo 1200mg vs Alpha Lipoic Acid (ALA) 1200mg; Test type: Superiority; p = 0.30, Mixed Models Analysis

5. Primary Outcome: Phase II: Mean Annual Growth of Geographic Atrophy (Fundus Autofluorescence) - Square Root of Area of GA (mm) - Adjusted
Description: as for outcome 4
Time Frame: 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Number analyzed (Participants) | 26 | 26
mm/year | 0.27 (0.04) | 0.32 (0.05)
Statistical Analysis 1: Comparison: Placebo 1200mg vs Alpha Lipoic Acid (ALA) 1200mg; Test type: Superiority; p = 0.14, Mixed Models Analysis

6. Secondary Outcome: Phase II: Mean Annual Change in Best-Corrected Visual Acuity (BCVA)
Description: Unit of Measure. Mean annual change in best-corrected visual acuity was calculated by taking the letter score at 18 months minus the baseline letter score. This value was then divided by 18 months and then multiplied by 12 months to get the mean annual change in visual acuity. Timepoints for the study were baseline, 0, 6, 12, and 18 months. The baseline and 18 month timepoints were used for the annualized calculations as noted below.
Time Frame: 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters/year
Arm/Group | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg
Number analyzed (Participants) | 26 | 26
letters/year | -3.8 (1.1) | -3.1 (1.12)
Statistical Analysis 1: Comparison: Placebo 1200mg vs Alpha Lipoic Acid (ALA) 1200mg; Test type: Superiority; p = 0.69, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Phase I: 15 Days; Phase II: 18 Months
Groups:
- Alpha Lipoic Acid (ALA) 1200 mg (Phase I): Phase I: All subjects recruited to the Phase I part will take escalating doses of alpha lipoic acid (ALA) open label. Each enrolled subject will take 600 mg of oral ALA once daily with a meal for 5 days. If well-tolerated, each subject will then take 800 mg of oral ALA once daily with a meal for 5 additional days. If 800 mg of oral ALA is well-tolerated, then subjects will then take 1200 mg of oral ALA once daily with a meal for 5 days.
- Alpha Lipoic Acid (ALA) 1200mg (Phase II): Phase II: All subjects in Phase II will be double blinded and randomized to either placebo or ALA. Each will take one 600 mg capsule of ALA (or placebo) once daily with a meal for 2 weeks and then increase to two 600 mg capsules of ALA (or placebo) once daily with a meal for the entire remainder of the 18 month period of the study.
Arm/Group | Alpha Lipoic Acid (ALA) 600 mg | Alpha Lipoic Acid (ALA) 800 mg | Alpha Lipoic Acid (ALA) 1200 mg (Phase I) | Placebo 1200mg | Alpha Lipoic Acid (ALA) 1200mg (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 1/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14 | 5/27 | 10/26
Other Adverse Events (participants affected / at risk) | 11/15 | 10/15 | 10/14 | 24/27 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha Lipoic Acid (ALA) 600 mg (N=15) | Alpha Lipoic Acid (ALA) 800 mg (N=15) | Alpha Lipoic Acid (ALA) 1200 mg (Phase I) (N=14) | Placebo 1200mg (N=27) | Alpha Lipoic Acid (ALA) 1200mg (Phase II) (N=26)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 2 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha Lipoic Acid (ALA) 600 mg (N=15) | Alpha Lipoic Acid (ALA) 800 mg (N=15) | Alpha Lipoic Acid (ALA) 1200 mg (Phase I) (N=14) | Placebo 1200mg (N=27) | Alpha Lipoic Acid (ALA) 1200mg (Phase II) (N=26)
Acid Reflux (Dyspepsia) (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 6 | 2
Loose Stools (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 7
Stomach Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 5
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Weakness (Asthenia) (General disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Leg (Muscle) Cramps (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Abnormal Urine Odor (Renal and urinary disorders) | 8 | 7 | 7 | 0 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Increased Urinary Frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hot Flashes (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Angle Closure Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 2
Blepharitis (Eye disorders) | 0 | 0 | 0 | 2 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 3
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 2
Macular Degeneration (Eye disorders) | 0 | 0 | 0 | 3 | 1
Retinal Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 2
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 4 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 6 | 7
Visual Disturbance (Eye disorders) | 0 | 0 | 0 | 3 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Giardiasis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 4 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 4 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 6 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 5
Back Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 3
Weight Decreased (Investigations) | 0 | 0 | 0 | 1 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
Hypertonic Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02613572/Prot_SAP_000.pdf